CLINICAL TRIAL: NCT03244670
Title: A Cohort Study on Incidence and Progression of Myopia in a Group of Medical Students
Brief Title: The Incidence and Progression of Myopia: Cohort Study
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Essilor International (Industry)
Responsible Party: Principal Investigator, Xiang Chen, Associate Professor, Sun Yat-sen University
Other Study IDs: TEX2017
Record Dates: First submitted 2017-08-07; First posted 2017-08-09 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Myopia
Keywords: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation study only, no specific intervention — Observation study only, no specific intervention

SUMMARY:
A cohort study on incidence and progression of myopia in a group of medical students

DETAILED DESCRIPTION:
A prospective cohort study to investigate the refractive error development, progression and their risk factors in young adult population comprises a group of medical students in China for two years

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subject, , willing to follow the protocol and able to read, comprehend and sign the informed consent form,
* Age between 17 and 23 years

Exclusion Criteria:

* Vulnerability of the subject,
* Participation in another study which might have an influence on vision or interfere with study assessments,
* Aphakic or pseudophakic (intraocular lens)
* Participants who are wearing ortho-K lenses, or undergone any kind of myopia control treatments or undergone refractive surgery.
* Any current or evolving pathology manifested in the eye or the appendages which might have an influence on vision, or interfere with study assessments (e.g. AMD, glaucoma…),
* Any previous ocular surgery which might have an influence on vision or interfere with study assessments (e.g. iridectomy, refractive surgery…),
* Any untreated and/or uncontrolled systemic condition which might have an influence on vision, or interfere with study assessments (e.g. uncontrolled diabetes, uncontrolled high blood pressure…),
* Any medical treatment or medication which might have an influence on vision or interfere with study assessments (e.g. antidepressants, drugs with atropinic effects…),

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: First-year medical college student from Zhongshan University
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-09-19 (Actual)

PRIMARY OUTCOMES:
refraction | Change from baseline for two years
  The participants will be measured for their refractive error by optometrist, and observe the rate of progression of myopia

CONTACTS AND LOCATIONS:
Overall Officials: Chen xiang, Principal Investigator — Associate Professor
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No